CLINICAL TRIAL: NCT06236087
Title: Assessing the Impact of Overdose Prevention Centers as a Polysubstance Use and Behavioral Health Intervention in New York City
Brief Title: Overdose Prevention Centers and Behavioral Health
Status: Not yet recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 23-01594; 23-A0-00-1010153 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Overdose
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aim 1 & 2 - Dataset: For Aims 1 and 2, an existing, de-identified dataset will be used for secondary analysis, including records for a maximum of 500 individuals.
  Aim 1 will use machine learning to identify sub-groups for whom OPC use is most and least protective of overdose risk. Identifying key intersectional groups across demographic (e.g., race/ethnicity, gender, and age), PSU factors (e.g., drug types and routes of administration), and socio-behavioral (e.g., mental health history, justice history, and homelessness) characteristics will inform targeted service delivery. Aim 2 will use epidemiological methods to estimate the association of OPC use with mental health services salient to PSU populations (e.g., hospitalization for depression, anxiety, and bipolar disorder). Measuring the association of OPC use with treated mental health outcomes for PSU-involved populations will foster an understanding of the impacts of OPCs on critical but unevaluated outcomes.
- Aim 3 - Harm Reduction Staff: For Aim 3, individuals employed at harm reduction programs in NYC will be enrolled for a one-time qualitative interview. Qualitative interviews will explore organizational (i.e., readiness, culture, and priorities), individual (i.e., attitudes and norms), and intervention (i.e., complexity and advantage) characteristics related to the integration of mental health and harm reduction services. Findings will inform efforts to scale ancillary mental health services high-risk PSU population.

SUMMARY:
The aims of this study are: (Aim 1) Identify sources of heterogeneous impacts of opioid prevention center (OPC) use on non-fatal and fatal overdose risk among individuals with histories of polysubstance use (PSU); (Aim 2) Estimate the impact of OPC use on treated psychiatric events among clients with histories of PSU, and; (Aim 3) Assess the barriers and facilitators of integrating mental health services into existing syringe service and OPC delivery models.

DETAILED DESCRIPTION:
Aims 1 and 2 of this study will use secondary data to identify sources of heterogeneous impacts of OPC use on fatal and nonfatal overdose risk (Aim 1) and estimate the impact of OPC use on treated psychiatric events among clients with histories of PSU (Aim 2). Aim 3 of this study will use qualitative interviews with harm reduction staff to assess barriers and facilitators of integrating mental health services into existing syringe service and OPC delivery models.

ELIGIBILITY:
Inclusion Criteria:

Aims 1 and 2:

* are 18 years of age or older;
* engaged in syringe service program and/or overdose prevention center services in New York City in the past 30 days before the date of enrollment;
* are able to complete assessments in English or Spanish;
* are competent to give written informed consent at the time of the interview;
* are able to provide informed consent;
* self-report use of illicit opioids (e.g., heroin, fentanyl), illicit stimulants (e.g., powder cocaine, crack, methamphetamine), counterfeit prescription pills (defined as prescription pills obtained through the illicit drug market) or any injection drug use in the past 30 days, and
* are able to participate for at least 6 months following enrollment.

Aim 3

* are 18 years of age or older;
* are employed by a harm reduction program;
* are able to complete assessments in English; and
* are able to provide informed consent.

Exclusion Criteria:

• Individuals not meeting the criteria detailed above for the respective Aims will not be eligible for participation in this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Aims 1 and 2 of this study will use secondary analysis of an existing de-identified, linked data set curated as part of an ongoing evaluation of the NYC overdose prevention centers. This dataset will include a total of 500 participants linked to NYC administrative health records. This de-identified data source will be accessed through the NYULH Center for Opioid Epidemiology and Policy (COEP). Should it be deemed necessary, a data use agreement will be established between the PI and NYULH/COEP to facilitate access to these de-identified data.
  Aim 3 of this study will recruit 30 individuals over age 18 who are currently employed by harm reduction programs for a one-time, qualitative interview.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Fatal Overdose | Up to Month 12
  Incidence of fatal overdose will be derived from overdose mortality data from the NYC Office of the Chief Medical Examiner.
Incidence of Non-Fatal Overdose | Up to Month 12
  Incidence of nonfatal overdose will be assessed using hospitalization and emergency department data from the NYC Regional Health Information Exchange (RHIO) and Statewide Research and Planning Cooperative System (SPARCS).
Incidence of Psychiatric Services Utilization | Up to Month 12
  Psychiatric services utilization will be assessed from SPARCS, RHIO, and NYS Medicaid.

CONTACTS AND LOCATIONS:
Overall Officials: Bennett Allen, PhD, MPA, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Bennett.Allen@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to bennett.allen@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.